CLINICAL TRIAL: NCT05578326
Title: Study of Trilaciclib and Lurbinectedin in Small Cell Lung Cancer
Brief Title: Study of Trilaciclib and Lurbinectidin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2117
Record Dates: First submitted 2022-09-23; First posted 2022-10-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer; Small-cell Lung Cancer
Keywords: Lurbinectedin; Trilaciclib; myelosuppression; neutropenia
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Neutropenia | interventions — trilaciclib; PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trilaciclib and Lurbinectedin (Experimental): Subjects with platinum refractory extensive stage small cell lung cancer receiving laciclib and Lurbinectedin
  Interventions: Drug: Trilaciclib; Drug: Lurbinectedin

INTERVENTIONS:
Drug: Trilaciclib — 240 mg/m2 intravenous, over 30 minutes at day 1 of each cycle
Drug: Lurbinectedin — 3.2 mg/m2, over 60 minutes at day 1 of each cycle

SUMMARY:
Lung cancer is by far the leading cause of cancer death among both men and women worldwide and the second most common cancer in terms of new cases. Small cell lung cancer (SCLC) is the deadliest form of lung cancer. The standard first-line treatment is the combination of carboplatin, etoposide, and atezolizumab. While response rates for this regimen are high (roughly 60%), the duration of response is short, typically 4 months. Following progression after the 1st line treatment of SCLC, there is no consensus regarding subsequent therapy. Lurbinectedin is FDA approved and is increasingly preferred in clinical practice. Toxicity was significant, but appeared favorable compared to historic results with topotecan, leading to the adoption of this therapy for second-line SCLC. The toxicity profile was dominated by myelosuppression.

This study investigates the effect of Trilaciclib on myelosuppression rate in subjects with platinum refractory extensive stage (ES)- SCLC receiving Lurbinectedin as well as the clinical synergy of Trilaciclib and Lurbinectedin combination.

ELIGIBILITY:
In order to participate in this study, a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Age ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Measurable disease according to RECIST v1.1 within 28 days prior to start of treatment.
* Previous treatment with a platinum agent, PD1 or PDL1 agent.

Exclusion Criteria:

* Active infection requiring systemic therapy.

  * Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
  * Treatment with any investigational drug within 4 weeks prior to start of treatment.
  * A known allergy or sensitivity to either study drug or its excipients.
  * Subject is receiving prohibited medications or treatments as listed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2027-12-25 (Estimated)

PRIMARY OUTCOMES:
The proportion of grade 4 neutropenia | Up to 21 days
  The proportion of subjects that experience grade 4 neutropenia as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 will be determined.
  CTCAE is descriptive terminology that can be used for Adverse Event (AE) grading and reporting. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
The duration of grade 4 neutropenia | Up to 21 days
  The median duration of subjects that experience grade 4 neutropenia as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 will be reported.

SECONDARY OUTCOMES:
The mean duration of grade 4 neutropenia | Up to 21 days
  The mean duration of grade 4 neutropenia in cycle 1 will be defined as the start of grade 4 neutropenia to the time of decreased grade as measured in days or censored at the time of death if a subject dies with Grade 4 neutropenia in Cycle 1.
The number of grade 3/4 anemia, grade 3/4 thrombocytopenia, and febrile neutropenia | Up to 8 months
  Toxicity will be evaluated, as the number of grade 3/4 anemia, grade 3/4 thrombocytopenia, and febrile neutropenia based on the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria, in any cycle (including cycle 1).
Use of secondary/reactive supportive measures | Up to 8 months
  To characterize use of secondary/reactive supportive measures any supportive measures such as Granulocyte colony-stimulating factor ( G-CSF) and erythropoietin stimulating agents (ESA) administration, red blood cell and platelet transfusion will be recorded.
Dose Intensity of Chemotherapy/ Number of chemotherapy dose reductions | Up to 8 months
  The dose Intensity of Chemotherapy/ Number of chemotherapy dose reductions will be defined as the ratio of the subjects who required chemotherapy dose reductions to all subjects who received study treatment.
Dose Intensity of Chemotherapy/ Number of chemotherapy cycles | Up to 8 months
  The dose Intensity of Chemotherapy/ Number of chemotherapy cycles will be defined as the median number of chemotherapy cycles among the subject who received study treatment.
Dose Intensity of Chemotherapy/ Number of chemotherapy delays | Up to 8 months
  The dose Intensity of Chemotherapy/ Number of chemotherapy delays will be defined as the median number of chemotherapy cycle delays dates among the subject who received study treatment.
Dose Intensity of Chemotherapy/ the total chemotherapy dose | Up to 8 months
  The dose Intensity of Chemotherapy/ the total chemotherapy dose will be defined as the median chemotherapy dose among the subject who received study treatment.
Overall Response Rate (ORR) | Up to 5 years
  To estimate the ORR, the proportion of subjects that respond (CR + PR) will be measured according to RESIST 1.1 will be calculated.
  RECIST: Radiographic response will be measured by RECIST, Response Evaluation Criteria In Solid Tumors Criteria, indicating if the subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Progression-free survival (PFS) | Up to 5 years
  PFS will be measured from the initiation of study therapy until progression per RECIST 1.1 or death of any cause or at last date of disease assessment if no progression is observed during the study period.
Overall survival (OS) | Up to 5 years
  OS will be measured from the initiation of therapy until death of any cause or censored at the last time known to be alive.
The kinetics of response | Up to 5 years
  The kinetics of response will be reported as tumor size over time for all patients, including the pace of progression from prior therapy.
QOL assessments FACT-L | Up to 5 years
  Scores from QOL assessments FACT-L version 4, from prior to study therapy through cycle 12 will be obtained, as described in the protocol.
  The FACT-L is a lung cancer specific subscale given at baseline, after each cycle and at end of treatment. Items are rated by patients on a Likert scale from 0 to 4. Higher scores represent better QOL.
QOL assessments FACT-An | Up to 5 years
  Scores from QOL assessments FACT-An version 4, from prior to study therapy through cycle 12 will be obtained, as described in the protocol.
  The FACT-An is an anemia specific subscale given at baseline, after each cycle and at end of treatment. Items are rated by patients on a Likert scale from 0 to 4. Higher scores represent better QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Lineberger Comprehensive Cancer Center at University of North Carolina Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials